CLINICAL TRIAL: NCT03940274
Title: Benefits of a Walk-Training Program on Cardiovascular Health in Individuals With Chronic Spinal Cord Injury (SCI)
Brief Title: Walk-Training Program for Individuals With Chronic Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00142564
Record Dates: First submitted 2019-04-04; First posted 2019-05-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injury
Keywords: Cardiovascular health; Walking training
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will undergo a walking program using a treadmill, a body-weight support system, and an assistive device.
  Interventions: Behavioral: walking training

INTERVENTIONS:
Behavioral: walking training — Participants will receive three sessions a week of BWSTT with assistive training device for 8 weeks; a total of 24 sessions. The duration of each training session will an hour. During walk-training, the participant will wear a harness which is attached to an overhead motorized lift to provide body-weight support and to prevent the risk of falling.

SUMMARY:
Cardiovascular disease (CVD) is the common leading cause of death among people with spinal cord injury (SCI) and occurs at an early age in people with SCI as compared to able-bodied people. The findings are consistent in demonstrating a high prevalence of CVD among people with SCI. Lack of physical activity and/or prolonged sitting which is observed in people with SCI due to impaired/loss of motor function is associated with increased risk factors of CVD. By doing this study, researchers hope to learn the effects of walking training on cardiovascular health among people with chronic SCI.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 60 years old, who have paraplegia (T1-L2) SCI, and who are scored less than 5 in Functional Independence Measure, Locomotion: Walk
* The onset of SCI must be one year or more at the beginning of the study
* Participants must not be participating in any other similar gait training activities
* Participants must have medical approval from their physician to participate in walk-training

Exclusion Criteria:

* Major Cardiovascular diseases
* Other neurological diseases
* Muscle spasticity (greater than 3 according to Ashworth scale)
* Severe orthopedic issues such as joint stiffness and fractures
* Osteoporosis (bone mineral density T-score less than - 2.5)[155]
* Inflammatory diseases or infections
* Open wound and pressure ulcer
* Pregnant women
* Cognitive or psychiatric disorders
* Uncontrolled autonomic dysreflexia; sudden increase in blood pressure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
The recruitment feasibility of an 8-week (3 sessions per week, 30 min per session) walk-training program in patients with chronic SCI. | From baseline to week 8
  Recruitment rate will be assessed by recording the number of participants who are screened for eligibility, those who are excluded because of eligibility criteria, and those who decline to participate in the study.
The perception feasibility of an 8-week (3 sessions per week, 30 min per session) walk-training program in patients with chronic SCI. | From baseline to week 8
  Information on perception will be acquired through a questionnaire that will be administered to participants at the end of walk-training program.
The compliance feasibility of an 8-week (3 sessions per week, 30 min per session) walk-training program in patients with chronic SCI. | From baseline to week 8
  Data on compliance rate will be documented during a period of training. The total number of completed sessions and incomplete sessions along with reasons for absence will be recorded throughout the study.
The retention feasibility of an 8-week (3 sessions per week, 30 min per session) walk-training program in patients with chronic SCI. | From baseline to week 8
  Data on retention will be obtained by recording the number of participants who drop out during the study along with their reasons.
The walking performance (walking time) feasibility of an 8-week walk-training program in patients with chronic SCI. | From baseline to week 8
  The time of walking (minutes) that a participant will be able to walk on a treadmill during each training session will be recorded.
The walking performance (treadmill walking speed) feasibility of an 8-week walk-training program in patients with chronic SCI. | From baseline to week 8
  The amount of treadmill speed (miles/hour) that a participant will be able to walk will be recorded during each training session.
The walking performance (number of stepping) feasibility of an 8-week walk-training program in patients with chronic SCI. | From baseline to week 8
  The number of stepping during each training session will be recorded using a step tracker.
Correlations between changes in four factors (muscle activity, cardiac autonomic function, spasticity, and lung capacity) and changes in heart rate after the walk-training program. | Change from baseline to week 8
  The resting heart rate will be measured during sitting position after 5 minutes rest. Exercise heart rate will be measured during a graded treadmill walking test with the same testing conditions pre- and post-training. The signal activity of four muscles in the lower limbs (biceps femoris, rectus femoris, gastrocnemius medialis, and tibialis anterior) will be measured using electromyography (EMG) system. The EMG recording will be obtained during walking on a treadmill. The average root-mean-square EMG for each muscle during gait cycle will be calculated. Cardiac autonomic function will be determined through power spectral of heart rate variability (HRV) using electrocardiography system. HRV frequency domain, including total power, low frequency (LF) and high frequency (HF) powers, and ratio of LF/HF, will be calculated and analyzed. Muscle spasticity for the lower extremities will be assessed through Modified Tardieu Scale. lung capacity will be measured through a spirometer.

SECONDARY OUTCOMES:
Changes in lipid profile after 8-week walk-training program. | Change from baseline to week 8
  For lipid profile, we will assess serum concentrations of total cholesterol, low density lipoprotein and high density lipoprotein using an enzymatic colorimetric assay.
Changes in the level of glycated hemoglobin (HbA1c) after 8-week walk-training program. | Change from baseline to week 8
  The level of HbA1c will be assessed using a device A1CNow+ System.
Changes in the level of pro-inflammatory markers after 8-week walk-training program. | Change from baseline to week 8
  For inflammatory markers, serum concentrations of C-reactive protein and interleukin-6 will be determined using an enzyme-linked immunosorbent assay.

OTHER OUTCOMES:
Changes in lower-limbs muscle strength after 8-week walk-training program. | Change from baseline to week 8
  Muscle strength will be evaluated using lower extremity motor score (LEMS), according to guidelines of the American Spinal Injury Association. LEMS is a manual muscle testing that assesses the strength of five key muscle groups of the lower extremities bilaterally: the hip flexors, knee extensors, ankle dorsiflexors, great toe extensors, and ankle plantarflexors. Each muscle group will be graded from 0 (absence of muscle contraction) to 5 (active movement with the full range of motion against full resistance). The total score of LEMS ranges from 0 to 50.
Changes in lower-limbs muscle spasticity after 8-week walk-training program. | Change from baseline to week 8
  Muscle spasticity will be assessed through the Modified Ashworth Scale (MAS). MAS is a subjective scale for clinical assessment of involuntary resistance to passive movement and, hence, muscle tone [166, 168]. An examiner will move the patient's limb through its full range of movement and will rate the amount of resistance felt. Resistance is rated based on a 6-point scale (grades 0, 1, 1+, 2, 3, 4), with lower scores indicating no spasticity and higher scores representing increasing resistance to passive movement.
Changes in muscle spasticity after 8-week walk-training program. | Change from baseline to week 8
  Muscle spasticity will subjectively be measured using the Penn Spasm Frequency Scale (PSFS). PSDS is a two components self-report questionnaire that assesses an individual's perception of spasticity frequency and severity. The first component is a 5-point scale assessing the frequency with which spasms occur ranging from "0 = No spasms" to "4 = Spontaneous spasms occurring more than ten times per hour. The second component is a 3-point scale assessing the severity of spasms ranging from "1 = Mild" to "3 = Severe". If an individual indicates that he/she has no spasms in the first component, the second component is not evaluated.
Changes in functional independence after 8-week walk-training program. | Change from baseline to week 8
  The Spinal Cord Independence Measure (SCIM) self-report version (SCIM-SR) will be utilized to evaluate the level of functional independence. This questionnaire contains 17 items, divided into three subscales: self-care (items 1-4), respiration and sphincter management (items 5-8), and mobility ability (items 9-17). The total score of SCM-SR ranges from 0 to100, which indicates the level of functional independence. The higher score represents a higher level of functional independence.
Changes in the level of depression, anxiety and stress after 8-week walk-training program. | Change from baseline to week 8
  Depression Anxiety Stress Scales-21 (DASS-21) will be used to determine the level of depression, anxiety, and stress. DASS-21 is a self-administered questionnaire that is designed to assess the negative emotional states of depression, anxiety, and stress over the past few weeks. It consists of three subscales with seven items in each subscale (total of 21 items). The response to each item is given on a 4-point Likert scale ranging from 0 = "Did not apply to me at all" to 3 = "Applied to me very much or most of the time". The score for each subscale is calculated by summing the scores for the relevant items. The low score indicates a normal level, whereas the high score indicates an extremely severe level of depression, anxiety, and stress.
Changes in health-related quality of life (HRQOL) after 8-week walk-training program. | Change from baseline to week 8
  Change in HRQOL will be assessed via the Short form-36 (SF-36). SF-36 is a self-reported, 36-items questionnaire that assesses eight domains of perceived HRQOL during the previous 4 weeks.[179, 180] The eight domains include physical functioning, role-physical functioning, bodily pain, general health, vitality, social functioning, role-emotional functioning, and mental health. The score for each domain ranges from 0-100. The higher score represents better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alajam RA, Alqahtanti AS, Frederick J, Liu W. The feasibility of an 8-Week walking training program using a novel assistive gait training device in individuals with spinal cord injury. Disabil Rehabil Assist Technol. 2022 Aug;17(6):658-667. doi: 10.1080/17483107.2020.1805801. Epub 2020 Aug 11. PMID 32780981

DOCUMENTS (1):
  • Study Protocol (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT03940274/Prot_000.pdf